CLINICAL TRIAL: NCT04630821
Title: Pilot Study of Utilizing Topical Sodium Hypochlorite to Ameliorate or Reduce Radiation Dermatitis
Brief Title: Utilizing Topical Sodium Hypochlorite to Ameliorate Radiation Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low participant accrual
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Paller, Chair, Department of Dermatology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AP09042019
Record Dates: First submitted 2020-11-11; First posted 2020-11-16 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Dilute Sodium Hypochlorite solution (Experimental): Subjects will be treated with the dilute bleach compresses daily (Monday through Friday) for the first 3 weeks of therapy. The bleach solution will be prepared and compresses applied for a 20 minute duration prior to radiation therapy. The compress can be applied within an hour of radiation therapy. Subjects will apply Aquaphor® ointment twice a day, once immediately after the radiation treatment and once in the evening. On days the experimental subjects do not receive radiation therapy, they will continue to moisturize their skin twice a day (AM and PM) with Aquaphor® ointment.
  Interventions: Other: Dilute Sodium Hypochlorite solution

INTERVENTIONS:
Other: Dilute Sodium Hypochlorite solution — Subjects will be treated with the dilute bleach compresses daily for the first 3 weeks of therapy.
  While these subjects are undergoing radiation therapy, they will be assessed weekly before the day's compress treatment by a physician investigator on the study team. Subjects will be evaluated and photographs will also be taken at study visits 1-3. The subjects will also complete a subject questionnaire addressing patient-reported outcomes at baseline and each weekly check-in during these two weeks. They will be also interviewed about ease of use and treatment tolerability. Subjects will complete interview questions at the end of the study to determine if they would continue the treatment and any obstacles or barriers.

SUMMARY:
The objective of the pilot study is to determine compliance, acceptability, and feasibility of using topical sodium hypochlorite to ameliorate or reduce radiation dermatitis, and to collect preliminary data and estimates for planning a larger efficacy study.

This 3-week single-arm pilot study will collect information on subject treatment compliance and feedback from subjects (and nurses/subject's treating oncologist) on the acceptability of the use of the treatment. We will also collect data on Common Terminology Criteria for Adverse Events and patient reported outcomes measured using the pain and pruritus PROMIS short-form tools and patient reported outcomes, measured using the Dermatology Life Quality Index (DLQI) tool.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Been diagnosed with head and neck cancer requiring radiation therapy or skin cancer requiring radiation treatment to the neck
* Are scheduled for a radiation therapy planning session (CT simulation)
* Have a scheduled radiation therapy start date within 1 to 2 weeks from the CT simulation
* Are able to comply with the study protocol

Exclusion Criteria:

* Patients who are pregnant, which may lead to discontinuation of radiation therapy
* Patients currently on immunotherapy
* Active or past history of inflammatory lesions in the radiation field that could interfere with assessment
* Patients who are undergoing re-irradiation to the head and neck
* Patients must not have any other condition or situation beyond those listed above which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the patient's participation in the study.
* Patients who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function are not eligible.
* Participation in other clinical trials that would alter the radiation dose typically utilized for definitive chemo and radiation therapy treatment of head and neck cancer.
* Use of other topical treatments on the skin in the treatment field. No other products are allowed except Aquaphor® ointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Compliance with compress application | 3 weeks
  Compliance will be measured as the proportion of subjects who complete 80% or more of the compresses. We will consider the study 'successful' if ≥ 80% of patients complete 80% or more of the compresses.
Occurrence of adverse events from compress application | 3 weeks
  The number of adverse events that occur in relation to the compress application will be tabulated during the course of the study.
Improvement in patient reported outcome measures | 3 weeks
  Patient reported outcome survey results will be scored prior to and after compress treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Department of Dermatology, Chair
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study results will be shared with our collaborative investigator at Boston Children's Hospital and Dana Farber/Harvard, Dr. Jennifer Huang, who is conducting a parallel adult study. This study will also inform our planned parallel studies with Dr. Huang in pediatric cancer patients undergoing radiation. Both sites will have access to each other's de-identified dataset once the appropriate Data Use Agreements are in place.
Supporting Information: CSR
Time Frame: at the end of data collection